CLINICAL TRIAL: NCT04552860
Title: Video Teleconference (VTC) Emotional Awareness and Expression Therapy (vEAET) for Older Veterans With Chronic Musculoskeletal Pain: An Initial, Uncontrolled Pilot Study
Brief Title: vEAET for Older Veterans With Chronic Musculoskeletal Pain Pilot
Acronym: vEAET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-000142
Record Dates: First submitted 2020-09-02; First posted 2020-09-17 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic Pain; Psychotherapy; Musculoskeletal Disease; Video Teleconference Delivered Therapy
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Video teleconference delivered Emotional Awareness and Expression Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Awareness and Expression Therapy (Experimental): Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Focus on emotions, writing about stress, assertiveness training, role playing new ways to handle relationships, and sharing feelings and experiences with others.
  Other Names: EAET

SUMMARY:
An uncontrolled pilot in which Veterans age 60-95 years with chronic musculoskeletal (MSK) pain will undergo Emotional Awareness and Expression Therapy (EAET) delivered over video teleconference (VTC; together vEAET). This study aims to obtain early implementation outcomes, as well as evaluate efficacy and estimated effect sizes.

DETAILED DESCRIPTION:
For this pilot, vEAET will be provided to outpatient Veterans age 60-95 years with chronic MSK pain in order to obtain early implementation and clinical outcomes (i.e. acceptability, feasibility, appropriateness, fidelity, and effectiveness). Each Veteran will be provided a VTC capable tablet and technological support from a research coordinator as a strategy to overcome technology based obstacles and obtain feasibility data. Veterans will receive one 90-minute individual session of vEAET plus eight 90-minute weekly group sessions of vEAET, all delivered over VTC to their homes. Assessments will be performed at baseline, posttreatment, and 2-month follow-up remotely using OutcomeMD (Los Angeles, CA), a HIPAA-compliant, VA-approved web-based platform. The entire study will be performed without any in-person visits.

ELIGIBILITY:
Inclusion Criteria:

• Eligible Veterans are age 60-95 years old and have had at least 3 months of musculoskeletal pain, including the following conditions most likely to benefit from psychotherapy based on previous research: low back, neck, leg, or pelvic pain; temporomandibular joint disorders; fibromyalgia; tension headaches; or any combination of these disorders.

Exclusion Criteria:

* Musculoskeletal conditions likely to respond surgical or pharmacologic treatment: hip or knee osteoarthritis, leg pain greater than back pain (to exclude radiculopathy), electromyography-confirmed "tunnel" syndrome (e.g., carpal tunnel syndrome), gout, neuralgias, migraine, and cluster headaches;
* Non-musculoskeletal pain conditions: autoimmune disease that typically generates pain (e.g., rheumatoid arthritis), cancer pain, sickle cell disease, burn pain, infection associated with pain, and cauda equina syndrome;
* The following conditions or circumstances: severe psychiatric disorder such as schizophrenia or bipolar I disorder not controlled with medications, active suicide or violence risk, active severe alcohol or substance use disorder, substantial cognitive impairment based on chart review, previously completed EAET, currently enrolled in another psychological treatment for chronic pain, currently in pain-related litigation or applying for pain-related compensation or compensation increase (e.g., VA service connection for chronic pain), unable to fluently read or converse in English, no internet access.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
The Satisfaction with Therapy and Therapist Scale-Revised | 8-Week Post-treatment
  Satisfaction with therapy subscale is the summation of six items, each scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction), yielding a total score between 6 and 30. Satisfaction with therapist subscale is the summation of six items, each scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction), yielding a total score between 6 and 30. Overall satisfaction is an additional single item scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction). The two subscales and the overall satisfaction item are each reported separately.
Credibility/Expectancy Questionnaire | Baseline
  Logical Credibility/Expectancy subscale is the average of four self report items, three of which are scored 1-9 (1 = not at all logical; 9 = very logical). A fourth Logical Credibility/Expectancy item reflects the percentage of functioning improvement participants think will occur. Feeling Credibility/Expectancy subscale is the average of four self report items, three of which are scored 1-9 (1 = not at all logical; 9 = very logical). A fourth Feeling Credibility/Expectancy item reflects the percentage of functioning improvement participants feel will occur. The two subscales are each reported separately.
Functional Assessment of Currently Employed Technology Scale (FACETS) | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  The summation of ten items related to ease of use of technology, each scored 1-6 (1 = never use a technology; 5 = easy/regular use of a technology), yielding a total score between 10 and 60.
Percent of Group Therapy Sessions Attended | 8 Weeks
  Number of sessions each participant attends divided by 8 sessions (total number of sessions available to attend).

SECONDARY OUTCOMES:
Anger Discomfort Scale | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  The summation of fifteen items related to Anger Discomfort, each scored 1-4 (1 = almost never; 5 = almost always), yielding a total score between 15 and 60. Three items are inverted scores.
Brief Pain Inventory (BPI) | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Average of four self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10.
Coping Strategies Questionnaire (CSQ) | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  The summation of fourteen items related to Coping Strategies, each scored 0-6 (0 = never do; 6 = always do), yielding a total score between 0 and 84. Two items are inverted scores.
Patient Reported Outcomes Measurement Information System (PROMIS)-Anxiety Short Form 7a | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Sum of seven self-report items assessing anxiety over the past 7 days. Items range from 1-5 (1 = never experiencing a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 7 and 35.
PROMIS-Depression Short Form 8a | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Sum of eight self-report items assessing depression and emotional distress over the past 7 days. Items range from 1-5 (1 = never feeling a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 8 and 40.
PROMIS-Global Health | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Global Physical health subscale is the summation of two items, each scored 1-5 (1 = excellent; 5 = poor), yielding a total score between 2 and 10. Global Mental health subscale is the summation of two items, each scored 1-5 (1 = excellent; 5 = poor), yielding a total score between 2 and 10. Health Perception & Social Roles subscale is the summation of two items, each scored 1-5 (1 = excellent; 5 = poor), yielding a total score between 2 and 10. The three subscales are each reported separately.
PROMIS-Pain Interference Short Form 8a | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Sum of eight self-report items assessing interference of pain with daily activities over the past 7 days. Items range from 1-5 (1 = no interference; 5 = maximum interference), yielding a total score between 8 and 40.
Property Association Task | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  One-hundred-thirty property-emotion pairs (e.g. frown-sadness) are assessed for the level of association between them on a scale of 0-6 (0 = not at all; 6 = extremely). Each pair represents a way of associating emotions to either interoception, behaviors, or situations (40 pairs each; 10 false pairs as controls). The three different association scores are summed up independently on a scale between 0 and 240. Answer reaction times are also collected.
PANAS Emotion Differentiation | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  The average of five self-report items assessing how much they current experience a certain emotional state. Items range from 0-100 (0 = Very slightly or not at all; 100 = Extremely).
Patient Global Impression of Change (PGIC) | 8-Week Post-treatment
  A single self report item assessing the Patient Global Impression of Change as a result of treatment. Items range from 1-7 (1 = No change (or condition has gotten worse); 7 = A great deal better and a considerable improvement that has made all the difference).
Social Connectedness Scale-Revised | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Sum of eight self-report items assessing feelings of Social Connectedness. Items range from 1-6 (1 = strongly agree/low connectedness; 5 = strongly disagree/high connectedness), yielding a total score between 8 and 48.
Survey of Pain Attitudes (SOPA) | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Sum of fourteen self-report items assessing the subject's attitude towards their pain. Items range from 0-4 (0 = this attitude is very untrue for me; 4 = this attitude is very true for me), yielding a total score between 0 and 56.
Test of Self-Conscious Affect 3-Short Version (TOSCA-3) | Change from Baseline, 8-Week Post-treatment, 2-Month Follow Up
  Forty-four self report items assess the likelihood of orientation towards feeling shame, detachment, guilt and externalization as reactions to eleven different scenarios. Items range from 1-5 (1 = not likely/low likelihood of reaction style; 5 = very likely/high likelihood of reaction style) and the four different reaction style scores are summed up independently on a scale between 11 and 55.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04552860/Prot_SAP_000.pdf